CLINICAL TRIAL: NCT06326528
Title: Short Term Outcome of SGLT2 Inhibitors on Patients Who Undergo Cardiac Surgery in Perioperative Period
Brief Title: SGLT2 Inhibitors and Perioperative Period
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nader Nabil, AssiutU, Assiut University
Other Study IDs: SGLT2 inhibitors
Record Dates: First submitted 2024-03-09; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Perioperative Complication
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGLT2 group: First group will receive SGLT2 (Dapaglifozin or Empagliflozin) inhibitors one month before surgery and three months after surgery.
  Interventions: Drug: SGLT2 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Dapagliflozin 10 mg or Empagliflozin 25mg
  Other Names: Dapagliflozin and Empagliflozin

SUMMARY:
The expanded use of SGLT2 inhibitors motivates us to assess the role of SGLT2 inhibitors in perioperative period on patients who will undergo cardiac surgery in Assiut University.

DETAILED DESCRIPTION:
With over 50 million cases of heart failure worldwide, heart failure is one of the most serious health issues facing humanity. Heart failure patients still have an extremely poor prognosis and quality of life, even with advancements in heart failure treatment. It continues to be the most common cause of hospitalization in elderly.

A substantial number of theories have been proposed to explain the beneficial effects of SGLT2 inhibitors. These include blood pressure lowering, increasing diuresis/natriuresis, improving cardiac energy metabolism, preventing inflammation, weight loss, improving glucose control, inhibiting the sympathetic nervous system, preventing adverse cardiac remodeling, preventing ischemia/reperfusion injury, inhibiting the cardiac Na/H exchanger inhibiting SGLT1, reducing hyperuricemia, increasing autophagy and lysosomal degradation, decreasing epicardial fat mass, increasing erythropoietin (EPO) levels, increasing circulating provascular progenitor cells, decreasing oxidative stress; and improving vascular function.

In addition to lowering blood sugar, several large trials also have demonstrated cardiovascular and renal benefits in patients with T2DM. Surprisingly, recent data also suggest that SGLT-2 inhibitors may improve cardiovascular and renal outcomes in patients without diabetes, leading to expanded indications for their use.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects with coronary artery disease or valvular heart disease referred to cardiac surgery

Exclusion Criteria:

1. Congenital heart disease.
2. Cardiomyopathy (EF>40%).
3. Sever renal impairment (eGFR>30).
4. COPD.
5. Marked obesity (BMI<35).
6. Previous cardiac surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac patients prepared for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference of cardiac function by speckle tracing between patients who will receive SGLT2 and patients who not. | six months
  We will measure cardiac function using speckle tracing method one month before cardiac surgery and three months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salma M Taha, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braunwald E. The war against heart failure: the Lancet lecture. Lancet. 2015 Feb 28;385(9970):812-24. doi: 10.1016/S0140-6736(14)61889-4. Epub 2014 Nov 16. PMID 25467564
- [Background] Verma S, McMurray JJV. SGLT2 inhibitors and mechanisms of cardiovascular benefit: a state-of-the-art review. Diabetologia. 2018 Oct;61(10):2108-2117. doi: 10.1007/s00125-018-4670-7. Epub 2018 Aug 22. PMID 30132036
- [Background] Staels B. Cardiovascular Protection by Sodium Glucose Cotransporter 2 Inhibitors: Potential Mechanisms. Am J Cardiol. 2017 Jul 1;120(1S):S28-S36. doi: 10.1016/j.amjcard.2017.05.013. Epub 2017 May 30. PMID 28606341
- [Background] Butler J, Handelsman Y, Bakris G, Verma S. Use of sodium-glucose co-transporter-2 inhibitors in patients with and without type 2 diabetes: implications for incident and prevalent heart failure. Eur J Heart Fail. 2020 Apr;22(4):604-617. doi: 10.1002/ejhf.1708. Epub 2020 Jan 11. PMID 31926059
- [Background] Filippatos TD, Liontos A, Papakitsou I, Elisaf MS. SGLT2 inhibitors and cardioprotection: a matter of debate and multiple hypotheses. Postgrad Med. 2019 Mar;131(2):82-88. doi: 10.1080/00325481.2019.1581971. PMID 30757937